CLINICAL TRIAL: NCT04856800
Title: Pre-meal Consumption of Whey in Gestational Diabetes Mellitus From Diagnosis to Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-10-72-326-20
Record Dates: First submitted 2021-03-23; First posted 2021-04-23 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2022-05

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Whey

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey (Experimental): Whey protein isolate WPI (Lacprodan® ISO.Water. from Arla Foods Ingredients). 20 g of whey protein will be ingested 30 min. prior to breakfast from diagnosis of GDM (around week 28) and until delivery.
  Interventions: Dietary Supplement: Whey
- Placebo (Placebo Comparator): The placebo will be ingested 30 min. prior to breakfast from diagnosis of GDM (around week 28) and until delivery.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Whey — 20 g protein of whey protein isolate WPI (Lacprodan® ISO.Water. from Arla Foods Ingredients)
  Arms: Whey
Dietary Supplement: Placebo — The placebo contains <1 kcal and 0 g protein
  Arms: Placebo

SUMMARY:
The main objective of the study is to investigate the metabolic effects of whey protein (whey protein isolate, WPI, (Lacprodan® ISO.Water. from Arla Foods Ingredients) compared with placebo when consumed by women with gestational diabetes mellitus (GDM) from diagnosis (around gestational week 28) to delivery. Any changes in substrate metabolism and energy expenditure using indirect calorimetry will also be investigated. Differences in hunger and satiety parameters as well as blood pressure and gestational weight gain will also be assessed. Furthermore, analysis on the glucose response when the women consume the intervention (whey or placebo) at home in their own environment 30 minutes before breakfast at time of diagnosis (earliest week 28) and week 36 (four days following each time point) will be made. The women will be monitored with continuous glucose monitors, activity monitors and all meals will be provided for two days following the study days in the laboratory. At delivery cord blood will be sampled for analysis on metabolic parameters and investigations on epigenetics/DNA methylations. Complications to the delivery, neonatal outcomes, anthropometrics of the child will also be assessed. Breast milk composition will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* GDM (OGTT level of blood glucose ≥ 9 mmol/L)
* Normal blood pressure
* Age > 18 years

Exclusion Criteria:

* Special dietary regimes > 1 month at time of inclusion e.g. ketogenic diet
* Daily intake of protein supplements
* Milk allergy or phenylketonuria
* Medication with effect on glucose metabolism e.g. steroids
* Do not speak or understand Danish
* Twin pregnancy
* PCOS
* PI finds the patient unfit (like mental illness, too nervous or other)
* Severe chronic illness
* Severe nausea/vomiting
* Non-breakfast eaters
* Celiac disease

The initiation of insulin treatment during the trial will not lead to exclusion from the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Maternal glycemic variability (GV) | 24 hours
  The Coefficient of Variation, power: n = 50
Maternal glycemic variability (GV) | 24 hours
  Interquartile range (IQR), power n = 40
Maternal glycemic variability (GV) | 24 hours
  Standard deviation (SD), power n = 18

SECONDARY OUTCOMES:
24 hours interstitial fluid glucose measures | 24 hours
  Continuous glucose monitoring
mean glucose | 24 hours
  Continuous glucose monitoring
maximum glucose | 24 hours
  Continuous glucose monitoring
Interstitial fluid glucose concentrations | 3 hours following breakfast
  Continuous glucose monitoring
Total energy expenditure | 24 hours
  Measured with a combined accelerometer and heart rate monitor, reported in kcal
Activity energy expenditure | 24 hours
  Measured with a combined accelerometer and heart rate monitor, reported in kcal
Activity count | 24 hours
  Measured with a combined accelerometer and heart rate monitor, reported in counts
Heart rate | 24 hours
  Measured with a combined accelerometer and heart rate monitor, reported in beats per minute
Resting energy expenditure (REE) (Resting Metabolic Rate) | Performed for 20 minutes
  Indirect calorimetry
Respiratory quotient (RQ) | Performed for 20 minutes
  Indirect calorimetry
Oxidation rates of lipid, carbohydrate and protein | Performed for 20 minutes
  Indirect calorimetry
Diet diary | 24 hours
  Total energy intake, composition of macronutrients
Self-reported appetite | 3,5 hours following intake of whey/placebo at diagnosis, week 32 and week 36
  Questionnaire: A numerical rating scale ranging from "not at all = 0" to "extremely = 10" will be used to assess Hunger, Fullness, Satiety, Desire, Prospective consumption (Quantity).
Body Mass Index | at diagnosis, week 32 and week 36
  weight and height will be combined to report BMI in kg/m^2
Gestational weight change | at diagnosis, week 32 and week 36
Medications | from diagnosis to delivery
  number of participants prescribed insulin, dose of insulin, time to insulin. Methyldopa, nifidipin or labetalol (medication to lower blood pressure)
Pregnancy data | from diagnosis to delivery
  Number of participants with hypertension, preeclampsia, maternal weight gain
Delivery data | at delivery
  Number of patients with cesarean section, shoulder dystocia, induction of labour
Non-targeted metabolomics will be performed on a sample of breast milk using Nuclear Magnetic Resonance | Day 1 postpartum
  Analysis generating metabolites from pathways on amino acids, peptides, carbohydrates and lipids measured in folds increase/decrease when comparing placebo with whey
Blood pressure | at diagnosis, week 32 and week 36
  Systolic and diastolic blood pressure
Concentration differences in Insulin like growth factor I (IGF-1) (mother) | at diagnosis, week 32 and week 36
Concentration differences in IGF-binding protein 3 (IGFBP-3) (mother) | at diagnosis, week 32 and week 36
Concentration differences in IGF-binding protein 1 (IGFBP-1) (mother) | at diagnosis, week 32 and week 36
Concentration differences in FGF-21 (mother) | at diagnosis, week 32 and week 36
Concentration differences in Leptin (mother) | at diagnosis, week 32 and week 36
Concentration differences in Adiponectin (mother) | at diagnosis, week 32 and week 36
Concentration differences in CRP (mother) | at diagnosis, week 32 and week 36
Concentration differences in Prolactin (mother) | at diagnosis, week 32 and week 36
Concentration differences in Cortisol (mother) | at diagnosis, week 32 and week 36
Concentration differences in Insulin (mother) | at diagnosis, week 32 and week 36
Concentration differences in Free Fatty Acids (mother) | at diagnosis, week 32 and week 36
Concentration differences in lactate (mother) | at diagnosis, week 32 and week 36
Concentration differences in grehlin (mother) | at diagnosis, week 32 and week 36
Concentration differences in inflammatory markers (IL-6, IL-10, IL-1α, IFN-γ, TNF-α)(mother) | at diagnosis, week 32 and week 36
Concentration differences in glucose independent peptide (GIP) (mother) | at diagnosis, week 32 and week 36
Concentration differences in glucagon like peptide 1 (GLP-1) (mother) | at diagnosis, week 32 and week 36
Concentration differences in glucagon (mother) | at diagnosis, week 32 and week 36
Concentration differences in c-peptide (mother) | at diagnosis, week 32 and week 36
Concentration differences in amino acids (AA) (mother) | at diagnosis, week 32 and week 36
Concentration differences in progesterone (mother) | at diagnosis, week 32 and week 36
Concentration differences in steroid hormone binding protein (SHBP) (mother) | at diagnosis, week 32 and week 36
Concentration differences in carboxy-terminal collagen crosslinks (CTx) (mother) | at diagnosis, week 32 and week 36
Concentration differences in osteocalcin (OCN) (mother) | at diagnosis, week 32 and week 36
Concentration differences in Pro-collagen I, N-term. pro-peptide (PINP) (mother) | at diagnosis, week 32 and week 36
Concentration differences in Human chorionic gonadotropin (HCG) (mother) | at diagnosis, week 32 and week 36
Concentration differences in CD163 (mother) | at diagnosis, week 32 and week 36
Concentration differences in estradiol (mother) | at diagnosis, week 32 and week 36
Concentration differences in hb1ac (mother) | at diagnosis, week 32 and week 36
Concentration differences in lipids (cholesterol, triglyceride) (mother) | at diagnosis, week 32 and week 36
Concentration differences in Insulin (cord blood, offspring) | at delivery
Concentration differences in c-peptide (cord blood, offspring) | at delivery
Concentration differences in glucagon (cord blood, offspring) | at delivery
Concentration differences in glucose (cord blood, offspring) | at delivery
Concentration differences in lactate (cord blood, offspring) | at delivery
Differences in pH (cord blood, offspring) | at delivery
  Measurement of acidity of the blood. Standard measurement performed on a sample of cord blood when a baby is delivered to evaluate possible oxygen deficiency during delivery.
non-targeted metabolomics analysis (cord blood, offspring) | at delivery
  Analysis generating metabolites from pathways on amino acids, peptides, carbohydrates, lipids and energy measured in folds rise/fall in when comparing placebo with whey
DNA methylations measured with 850K-Illumina Infinium assay. | at delivery
  Differentially methylated sites or regions associated with the intervention will be assessed.
RNA-Seq transcriptome profiling | at delivery
  Up and down-regulated genes associated with the intervention will be assessed
Body fat (offspring) | at delivery
  Sum of skinfolds measured with a caliper
Birth weight (offspring) | at delivery
Head circumference (offspring) | at delivery
abdominal circumference (offspring) | at delivery
Length (offspring) | at delivery
Number of infants with icterus | through hospital admission immediately after delivery
Apgar-score | at delivery
  Apgar score, range from 0-10, with the higher score the better outcome.
number of patients needing early feeding | through hospital admission immediately after delivery
Number of days admitted immediately after delivery | through hospital admission immediately after delivery
Number of infants with hypoglycemia | at delivery
Weight of placenta | at delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Medicinsk forskningslaboratorium for Diabetes og Hormonsygdomme og Steno Diabetes Center Aarhus (M-lab), Aarhus universitetshospital, Aarhus, Denmark